CLINICAL TRIAL: NCT04106635
Title: Effect of Pressure to Left Paratracheal Esophagus During the Insertion of Laryngeal Mask Airway
Brief Title: Effect of Paratracheal Esophagus Pressure on the Insertion of Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MED-INT-19-361
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: General Anesthesia; Pulmonary Aspiration
Keywords: Laryngeal mask airway; Paratracheal esophageal pressure; Cricoid pressure

STUDY DESIGN:
Intervention Model Description: Randomized double blinded clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The group assignments were sealed in opaque envelopes by a research assistant not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PP group (Experimental): During the induction of anesthesia, left paratracheal pressure is applied by 30N force with thumb after confirmation of the location of the esophagus using ultrasound.
  Interventions: Procedure: Paratracheal pressure
- CP group (Active Comparator): During the induction of anesthesia, cricoid pressure is applied by 30N force with three finger.
  Interventions: Procedure: Cricoid pressure

INTERVENTIONS:
Procedure: Paratracheal pressure — To apply paratracheal pressure, the thumb was placed over the left side of the trachea cephalad to the clavicle and medial to the sternocleidomastoid muscle.
  Arms: PP group
Procedure: Cricoid pressure — To apply cricoid pressure, the cricoid cartilage is compressed by 30N force with a single-handed three finger maneuvre towards the vertebral bodies.
  Arms: CP group

SUMMARY:
Laryngeal mask airway is inserted into the oral cavity and seals the upper esophagus and the surrounding tissue, effectively securing airway. Laryngeal mask airway has been widely adopted in the clinical practice.

On the other hand, cricoid pressure has been used to reduce the risk of pulmonary aspiration of gastric contents during induction of general anesthesia. However, cricoid pressure might impede placement of the laryngeal mask airway, thereby preventing effective ventilation.

Recently, left paratracheal pressure was introduced as an alternative to cricoid pressure and reported to be more effective than cricoid pressure in the prevention of gastric air insufflation during positive-pressure ventilation by facemask. Since this method compresses low left paratracheal level, it may affect the successful insertion of laryngeal mask airway.

In this study, the investigators aimed to evaluate the effect of paratracheal esophagus pressure on the insertion of laryngeal mask airway compare to conventional cricoid pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing surgery under general anesthesia where supraglottic airway management will be appropriate
* American Society of Anesthesiologists Classification 1-2

Exclusion Criteria:

* Body mass index > 35 kg/m2
* High risk of regurgitation (hiatus hernia, gastro-esophageal reflux disease, non-fasting status)
* Criteria for difficult airway (limitation of mouth opening/neck extension, Mallampati class IV),

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
The success rate of device insertion | During induction of anesthesia, an average of 60 seconds
  Successful insertion of laryngeal mask airway in a maximum of three attempts

SECONDARY OUTCOMES:
The grade of fiberoptic bronchoscopic view | During induction of anesthesia, an average of 5 minutes
  The fiberoptic bronchoscopic view is defined as Grade 1, larynx only seen; Grade 2, larynx and epiglottis posterior surface seen; Grade 3, larynx, and epiglottis tip or anterior surface seen-visual obstruction of epiglottis to larynx: < 50%; Grade 4, epiglottis down-folded, and its anterior surface seen-visual obstruction of epiglottis to larynx: > 50%; Grade 5, epiglottis downfolded and larynx cannot be seen directly.
The time for successful insertion of the device | : During induction of anesthesia, an average of 60 seconds
  The total time is measured from the removal of the face mask until bilateral chest rise with the first capnogram upstroke.
Peak inspiratory pressure | At 5 minute after insertion of laryngeal mask airway
  Peak inspiratory pressure is recorded from mechanical ventilator.
The ease of insertion of device | During induction of anesthesia, an average of 60 seconds
  The ease of placement was assessed using a subjective scale of 1-4 (1= no resistance, 2 = moderate resistance, 3 = high resistance, 4 = inability to place the device
The number of attempts at insertion of device | During induction of anesthesia, an average of 60 seconds
  The number of attempts for successful insertion of laryngeal mask airway
Success rate in first attempt | : During induction of anesthesia, an average of 60 seconds
  Successful insertion of laryngeal mask airway in a first attempt
Incidence of intraoperative complications | During the surgery, an average of 2 hours after anesthesia induction
  Intraoperative complications including coughing, laryngospasm, bronchospasm, hypoxia (SpO2 < 90%), regurgitation, aspiration, blood staining of the device.
Incidence of postoperative complications | An average of 2 hours after extubation
  Postoperative complications including sore throat, hoarseness/dysphonia, jaw, neck or ear pain, persistent cough, tachypnea, stridor, hypoxia (SpO2 < 90%), nausea and vomiting.
The presence of gastric air insufflation after induction of anesthesia | During induction of anesthesia, an average of 5 minutes
  The presence of gastric air insufflation is defined as an increase in antral cross-sectional area and/or presence of air artifacts in the antrum (comet tail, posterior acoustic shadow) confirmed by ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou university hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No